CLINICAL TRIAL: NCT05733143
Title: A Cross-sectional Study Using Cardio-pulmonary Exercise Stress Testing to Understand Physiological Differences in t2-biomarker Low Severe Asthma
Brief Title: Using Exercise-testing to Explore Patient Differences in Severe Asthma
Status: Active, not recruiting | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Liam Heaney, Professor of Respiratory Medicine, Queen's University, Belfast
Other Study IDs: B22/23; 320351 (Other: IRAS ID)
Record Dates: First submitted 2023-01-31; First posted 2023-02-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: asthma; Cardiopulmonary exercise stress testing
MeSH Terms: conditions — Asthma | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Haematology [5ml] (haemoglobin, haematocrit, platelet count, red blood cell count, white blood cell count, percent and absolute differential count.
  Samples for Biomarkers: The following will be collected on the day of Cardiopulmonary exercise stress testing for exploration of biomarkers and stored for future research. These biomarkers can include, but are not limited to, plasma biomarkers related to asthmatic airway inflammation, corticosteroid signalling and putative inflammatory pathways in severe asthma.
  * Plasma: 10 ml EDTA collection tube resulting in ~5 ml plasma stored as 0.5 ml aliquots for plasma measures of biomarkers related to asthmatic airway inflammation, corticosteroid signalling and putative inflammatory pathways in severe asthma
  * Urine sample: urinary eicosanoids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Symptom high/T2-biomarker low (20 participants): [ACQ≥ 1.5 FeNO<20 ppb AND blood eosinophil count<150 cells/µL]. During the study visit patients will undergo the following; COVID Lateral flow test (24 and 48 hours prior to assessment visit), Informed consent, Medical history and baseline demographics, vital Signs measurements, Weight/Height/BMI, Medication review, Concomitant medication check including technique, medical adherence, and self-management plan, Physical examination, Urine pregnancy test (If relevant), HADS score for depression, HADS score for anxiety, ACQ-5, Mini-AQLQ (QoL), St Georges Respiratory Questionnaire (SGRQ), Nijmegen hyperventilation score, BORG score, WHO Physical Global Activity Questionnaire (GPAQ), Haematology (FBC), Bio-banked samples: EDTA and urine(Eicosanoids), Spirometry, FeNO, Exercise test (CPEST) At 6 month follow up, in routine clinical care, participants will complete the same assessments. They will not be required to provide samples for biobanking or perform a repeat CPEST.
  Interventions: Other: cardiopulmonary exercise stress test (CPEST)
- Symptom low/T2-biomarker high (20 participants): [ACQ<1.5 AND FeNO≥20 ppb AND blood eosinophil count≥150 cells/µL] During the study visit patients will undergo the following; COVID Lateral flow test (24 and 48 hours prior to assessment visit), Informed consent, Medical history and baseline demographics, vital Signs measurements, Weight/Height/BMI, Medication review, Concomitant medication check including technique, medical adherence, and self-management plan, Physical examination, Urine pregnancy test (If relevant), HADS score for depression, HADS score for anxiety, ACQ-5, Mini-AQLQ (QoL), St Georges Respiratory Questionnaire (SGRQ), Nijmegen hyperventilation score, BORG score, WHO Physical Global Activity Questionnaire (GPAQ), Haematology (FBC), Bio-banked samples: EDTA and urine(Eicosanoids), Spirometry, FeNO, Exercise test (CPEST) At 6 month follow up, in routine clinical care, participants will complete the same assessments. They will not be required to provide samples for biobanking or perform a repeat CPEST.
  Interventions: Other: cardiopulmonary exercise stress test (CPEST)
- Symptom low/T2-biomarker low (12 participants): [ACQ<1.5 AND FeNO<20 ppb AND blood eosinophil count<150 cells/µL] During the study visit patients will undergo the following; COVID Lateral flow test (24 and 48 hours prior to assessment visit), Informed consent, Medical history and baseline demographics, vital Signs measurements, Weight/Height/BMI, Medication review, Concomitant medication check including technique, medical adherence, and self-management plan, Physical examination, Urine pregnancy test (If relevant), HADS score for depression, HADS score for anxiety, ACQ-5, Mini-AQLQ (QoL), St Georges Respiratory Questionnaire (SGRQ), Nijmegen hyperventilation score, BORG score, WHO Physical Global Activity Questionnaire (GPAQ), Haematology (FBC), Bio-banked samples: EDTA and urine(Eicosanoids), Spirometry, FeNO, Exercise test (CPEST) At 6 month follow up, in routine clinical care, participants will complete the same assessments. They will not be required to provide samples for biobanking or perform a repeat CPEST.
  Interventions: Other: cardiopulmonary exercise stress test (CPEST)
- Symptom high/T2-biomarker high (12 participants): [ACQ≥ 1.5 AND FeNO≥20 ppb AND blood eosinophil count≥150 cells/µL] During the study visit patients will undergo the following; COVID Lateral flow test (24 and 48 hours prior to assessment visit), Informed consent, Medical history and baseline demographics, vital Signs measurements, Weight/Height/BMI, Medication review, Concomitant medication check including technique, medical adherence, and self-management plan, Physical examination, Urine pregnancy test (If relevant), HADS score for depression, HADS score for anxiety, ACQ-5, Mini-AQLQ (QoL), St Georges Respiratory Questionnaire (SGRQ), Nijmegen hyperventilation score, BORG score, WHO Physical Global Activity Questionnaire (GPAQ), Haematology (FBC), Bio-banked samples: EDTA and urine(Eicosanoids), Spirometry, FeNO, Exercise test (CPEST) At 6 month follow up, in routine clinical care, participants will complete the same assessments. They will not be required to provide samples for biobanking or perform a repeat CPEST.
  Interventions: Other: cardiopulmonary exercise stress test (CPEST)

INTERVENTIONS:
Other: cardiopulmonary exercise stress test (CPEST) — The study is observational and purely exploratory. We will utilise cardiopulmonary exercise stress testing to assess levels of fitness and causes for symptoms in proposed groups.

SUMMARY:
The goal of this observational pilot study is to use exercise-testing to assess patients with severe asthma who have high levels of breathlessness and compare them to other groups of patients with low levels of breathlessness. We will compare the background and overall fitness levels in all groups. This may provide new knowledge to why these patients remain breathless despite being on treatment with low levels of inflammation.

The main question we aim to answer is:

"How are these patients different compared to patients who respond to treatment?" We will look at reasons why patients with low levels of inflammation in their lungs are still breathless despite being on treatment.

Participants will be required to take part in a 6-month study were they will firstly attend a "study visit" and a 6 month follow up.

At the study visit participants will be consented and required to:

* Complete questionnaires on their symptoms
* Provide information on their background
* Undergo a physical examination
* Provide blood and urine samples for specific testing for asthma and future investigations
* Perform breathing tests
* Undergo an exercise-test on a treadmill

During this study, researchers will compare this group will to participants who are similar but whose symptoms respond to treatment. We will also look at other groups of asthma patients who have who have different levels of inflammation in their lungs to see if there are any differences. We predict, these patients will have a different background and features to those whose symptoms respond to treatment.

DETAILED DESCRIPTION:
Introduction:

Asthma affects approximately 300 million people globally with a prevalence as high as 15% and was estimated to be the cause of 461,000 deaths in 2019. Asthma has a higher disability adjusted life-years per 100,000 population than diabetes and breast cancer, with much of this excess disability reported in the 10-20% of asthmatics who have challenging disease control. Traditionally, asthma management guidelines advocate a stepwise approach incrementally increasing CS along with other adjunctive therapies to achieve symptom control whilst reducing exacerbations. Current guidelines also recommend reducing CS after 3 months when optimal control is achieved. For many patients, this strategy works well, but in patients with severe asthma, symptoms often persist despite being on maximal treatment. At present, there is no standardised objective assessment tool when assessing patients with severe asthma who remain highly symptomatic.

Pathophysiology:

Asthma is underpinned by type-2 (T2) cytokine driven eosinophilic inflammation, with well-defined key inflammatory cytokines (interleukins (IL) -4, IL-5 and IL-13), and it is this inflammatory process which responds to CS treatment (6). All currently available new biologic therapies specifically target the T2-cytokine axis (IL-5 [mepolizumab, benralizumab and reslizumab], IL-4/13 [IL4R blockade -dupilumab]. Other drugs target upstream pathways by inhibiting epithelial alarmins [IL-33 and thymic stromal lymphopoietin (TSLP - Tezepelumab, currently not approved). These multiple new biologic treatments are primarily aimed at reducing acute asthma exacerbations and oral CS exposure. This inflammatory process can be assessed in the clinic using routinely measured biomarkers, blood eosinophil count (IL-5) and fractional exhaled nitric oxide (FeNO [IL-13]). Subsequently, patients are considered "T2-biomarker low" when FeNO <20 and blood eosinophils <150 (T2-biomarker low). Additional CS treatment or currently available biologic therapy has not proven to have any therapeutic benefit in patients who are T2 biomarker low. Furthermore, it is increasingly clinically recognised that symptoms of breathlessness and wheeze in this severe asthma population are often due to extra pulmonary co-morbidities (obesity and anxiety/depression). Treating these symptoms with CS or biologic therapy results in both treatment failure and the inappropriate continuation of high dose CS treatment leading to multiple side-effects.

Rationale for the study:

A particular patient sub-group (highly symptomatic with absence of eosinophilic airway inflammation) are sometimes referred to as having 'discordant disease' (dissociation between symptoms and T2 biomarkers) and represent a significant unmet clinical need. This T2-biomarker low population are predominantly female with a high prevalence of obesity and mood disturbance (anxiety/depression), suggesting that extra-pulmonary factors significantly influence symptoms in this sub-group of severe asthmatic female patients. Other data supports these observations, including a previous cluster analysis, which highlighted a spectrum of phenotypes existing within severe asthma and notably, this "obese non-eosinophilic" (T2 biomarker low) predominantly female group of patients was clearly identified. No specific treatment targets this group and other mechanisms are likely to be involved in persisting symptoms. A key step in assessing and managing this group is to develop a systematic process for identifying the reasons for persistent symptoms, including those not specifically related to asthma, and we believe CPEST testing is ideally suited for this purpose.

Rationale for Cardiopulmonary exercise stress testing One clinically useful tool in determining the mechanism of symptoms in patients with severe asthma is CPEST. CPEST can be used to identify contributory factors, other than asthma, for example hyperventilation, breathing pattern disorder, inducible laryngeal obstruction, ventilatory limitation due to fixed airflow obstruction, and physical deconditioning. A previous retrospective study assessing the use of CPEST in an unselected difficult asthma population identified multiple non-pulmonary mechanisms for physiological limitations as well as patients with normal CPEST despite self-reported high symptom burden. They found CPEST can be used to target treatment more appropriately including reduction of high dose CS therapy. However, this study did not relate symptoms to underlying T2-biomarkers, which were not routinely measured at that time, which is a critical novel component of this study.

At present, standard care in asthma is not assessment driven or based on objective testing through modalities such as CPEST. We will study patients with "discordant" disease (T2-biomarker and symptoms not aligned) and "concordant" disease (T2-biomarker and symptoms are aligned). Biomarker low will be defined as per GINA guidelines as (FeNO<20 ppb AND blood eosinophil count<150 cells/µL) and symptom low will defined as ACQ <1.5. 64 patients will be recruited to this trial and sub-grouped depending on T2 biology and symptoms, as below:

Discordant disease (n= 40) A) Symptom high/T2-biomarker low (20 participants) B) Symptom low/T2-biomarker high (20 participants)

Concordant disease (n= 24) C) Symptom low/T2-biomarker low (12 participants) D) Symptom high/T2-biomarker high (12 participants)

Study Aim:

To assess the key demographic, clinical and physiological differences in these distinct patient groups with severe asthma to define mechanisms of persistent breathlessness and exertional limitation in T2-biomarker low patients.

Hypothesis:

We hypothesise that CPEST will precisely determine the mechanism of persistent breathlessness and exertional limitation in symptom high (ACQ ≥ 1.5) but T2-biomarker low (FeNO<20 ppb AND blood eosinophil count<150 cells/µL) patients, allowing better targeting of intervention strategies to improve symptom burden in this sub-group.

OBJECTIVES AND OUTCOME MEASURES:

To describe maximal exercise tolerance and limiting factors at peak exercise in distinct patient groups with severe asthma - the following physiological parameters will be recorded (Findings are not limited to these parameters):

* Peak oxygen content/VO2 max (PVO2)
* Anaerobic threshold (AT)
* Maximum heart rate (HRmax)
* Blood pressure response (BP)
* Inspiratory flow-volume loop parameters,
* Post exercise spirometry
* Peak exercise O2 pulse
* Ventilatory reserve (% of MVV)
* SpO2 (%) at peak
* End-tidal CO2
* Ventilatory equivalent for carbon dioxide and oxygen (Ve/VCO2 and Ve/VO2) at anaerobic threshold R
* Resting/peak respiratory exchange ratio

We will also relate the above physiological measures to the below routinely measured asthma parameters and measures of physical activity:

Symptom scores (ACQ-5, BORG score) Quality of life scores/assessments (Mini-asthma quality of life questionnaire [mini-AQLQ] and St Georges Respiratory Questionnaire [SGRQ]) Levels of anxiety (Hospital Anxiety-Depression score [HADS]) Levels of depression (HADS score) Hyperventilation (Nijmegen Questionnaire) Short acting beta-2 agonist usage (SABA usage) [Dispensing records] Biomarker levels (blood Eos and FeNO) WHO Physical Global Activity Questionnaire (GPAQ)

Exercise test will be reviewed by a cardiopulmonary test expert blinded to biomarker profile to determine clinical diagnosis caused exertional limitation based on exercise test data.

Exploratory analysis:

The CPEST results will be available to clinic staff (as would be in normal clinical practice) and a treatment plan addressing any factors will be determined at the severe asthma multi-disciplinary team (MDT) meeting. Referrals may be made to MDT members including physiotherapy, speech-and-language therapy and clinical psychology in keeping with standard care in clinical practice.

The patients in this study will be followed up in routine care after 6 months to identify outcomes as below:

* Symptom scores (ACQ5, BORG score)
* Quality of life score/assessments (Mini-asthma quality of life questionnaire [mini-AQLQ] and St Georges Respiratory Questionnaire [SGRQ])
* Levels of anxiety (HADS score)
* Levels of depression (HADS score)
* Level of hyperventilation (Nijmegen Questionnaire)
* Perception of physical activity (WHO Physical Global Activity Questionnaire)
* SABA usage (Dispensing records [within 1 year])
* Dose of CS at study endpoint
* Requirement for rescue course of prednisolone or hospital admission for asthma at time of follow up
* Proportion of patients on OCS at study end
* Changes in lung function (between study completion and 6 month follow up)
* Biomarker levels (blood Eosinophils and FeNO)

The observational follow up review may provide useful pilot data to allow powering of a formal randomised control trial of multi-disciplinary intervention in this biomarker-low, symptom high population.

STUDY SETTING This is a UK single centre study at the tertiary care difficult asthma service at Belfast Health & Social Care Trust. CPEST will be performed at the Clinical Research Facility on the Belfast City Hospital Site (Wellcome-Wolfson Institute for Experimental Medicine) with the presence of primary investigator/delegate and CPEST physiologist.

ELIGIBILITY:
Inclusion Criteria

All participating patients will be attending the Regional Severe Asthma Service of Belfast Trust and will be:

1. Age ≥ 18 and ≤ 80 years at screening visit
2. Able and willing to provide written informed consent and to comply with the study protocol
3. Severe asthma confirmed after assessment by an asthma specialist as per GINA guidelines (1)
4. Diagnosed with asthma at least 12 months prior to screening and on GINA Step 4/5 treatment including those who are on biologic therapy
5. On optimal medical management as determined by clinician

Exclusion criteria

Exclusion criteria will be:

1. Any absolute contraindication to CPEST (Acute myocardial infarction (3-5 days), unstable angina uncontrolled arrhythmia causing symptoms or haemodynamic compromise, syncope, active endocarditis, acute myocarditis/pericarditis, symptomatic severe aortic stenosis, uncontrolled heart failure, suspected dissecting or leaking aortic aneurysm, uncontrolled asthma, arterial desaturation at rest on room air <85%) (15)
2. Acute exacerbation requiring oral corticosteroids in previous 4 weeks before first visit
3. History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the participant's full participation in the study, in the opinion of the investigator
4. Treatment with an investigational agent within 30 days of assessment (or five half-lives of the investigational agent, whichever is longer)
5. Female participants who are pregnant or lactating
6. Other clinically significant medical disease or uncontrolled concomitant disease despite treatment that is likely, in the opinion of the investigator, to impact the patient's ability to participate in the study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will aim to look at and sample phenotypically different groups of asthma patients who are symptom high and low with with either low or high biomarkers.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
OBJECTIVES AND OUTCOME MEASURES | 6 months
  The outcomes of this study are purely exploratory. We will describe maximal exercise tolerance and limiting factors at peak exercise in distinct patient groups with severe asthma using the physiological parameters derived from CPEST.

OTHER OUTCOMES:
EXPLORATORY ANALYSIS | 6 MONTHS
  CPEST results will be available to clinic staff (as would be in normal clinical practice) and a treatment plan addressing any factors will be determined at the severe asthma multi-disciplinary team (MDT) meeting. Referrals may be made to MDT members including physiotherapy, speech-and-language therapy and clinical psychology in keeping with standard care in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Liam G Heaney, MD, Principal Investigator — Queens University Belfast
Locations (1):
- Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All patient data will be anonymised during this study. Patients will have the option to consent for the use of their anonymised data in future work. As per normal practices, data will be stored for up to 15 years

REFERENCES:
- [Background] McNicholl DM, Megarry J, McGarvey LP, Riley MS, Heaney LG. The utility of cardiopulmonary exercise testing in difficult asthma. Chest. 2011 May;139(5):1117-1123. doi: 10.1378/chest.10-2321. Epub 2011 Feb 3. PMID 21292756